CLINICAL TRIAL: NCT02810080
Title: FiO2 Closed Loop Control Using the ZOLL 731 Series Ventilator
Brief Title: FiO2 Closed Loop Control Ventilation
Acronym: CLC
Status: Completed | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9703
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2023-04

CONDITIONS: Wounds and Injuries; Respiratory Failure
MeSH Terms: conditions — Wounds and Injuries; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (2):
- Closed Loop Control Ventilation (Experimental): automatic adjustment of the ZOLL 731 ventilator FiO2 by the closed loop control software
  Interventions: Device: Closed Loop Control Ventilation
- Manual Control Ventilation (Active Comparator): manual adjustment of the ZOLL 731 ventilator FiO2 by the treatment team based on physician order
  Interventions: Device: Manual Control Ventilation

INTERVENTIONS:
Device: Closed Loop Control Ventilation — Closed loop control ventilation using ZOLL 731 ventilator with physiologic closed-loop control software
  Arms: Closed Loop Control Ventilation
Device: Manual Control Ventilation — Manual control ventilation using ZOLL 731 ventilator
  Arms: Manual Control Ventilation

SUMMARY:
A randomized, multi-center trial involving critically-ill patients comparing conventional, manual control of inspired oxygen (FiO2) within a target range, with a computer-controlled, closed-loop FiO2 delivery using a continuous ventilator.

DETAILED DESCRIPTION:
The trial will use a proportional-integral-derivative (PID) type controller for automatic adjustment of FiO2 to maintain the SpO2 within a target range, based on continuous use of pulse oximetry. Intubated subjects will be randomized to either manual control of FiO2 or closed-loop control of FiO2, during a 12-hour period. The PCLC is designed to respond to acute hypoxemia (SpO2 <88%) within seconds while preventing hypoxemia and minimizing exposure to excessive inspired oxygen levels.

ELIGIBILITY:
Inclusion Criteria:

* The subject's legally authorized representative will provide signed and dated informed consent.
* Age 18 - 65, inclusive.
* Admission to a surgical or neurosurgical intensive care unit following traumatic injury or acute surgical illness
* Requirement for endotracheal intubation
* Requirement for mechanical ventilation
* Patient is currently receiving inspired oxygen concentration (FiO2) >=40%

Exclusion Criteria:

* Age under 18 or over 65
* Isolated or severe head injury (Glasgow Coma Scale = 6 or less) with expected survival less than 24 hours
* Brain death
* Anticipated survival less than 48 hours
* Pregnant female
* Patient in whom a pulse oximeter cannot detect a reliable signal due to hypotension, hypothermia, or other injury
* Known carbon monoxide poisoning
* Uncontrolled diabetic
* Patient who is unable to maintain SpO2 level of 88% at an FiO2 of 100% due to their medical condition. (NOTE: Being in the trial would impose no additional risk to a patient who presents with this condition however, data from a patient presenting with this pathophysiology would not provide insight into the performance of the controller as it would simply maintain that patient on an FiO2 of 100%.)
* Patient with chronic hypercarbia.
* Patient where a physician believes that FiO2 PCLC could be detrimental to the management of the patient.
* Prisoner
* SpO2 to SaO2 difference >4%
* Patient with core temperature <35 C

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-12; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Closed Loop Control Ventilation | Manual Control Ventilation
Started | 104 | 102
Completed | 97 | 98
Not Completed | 7 | 4
Not completed — Adverse Event | 3 | 0
Not completed — Death | 0 | 2
Not completed — Physician Decision | 4 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Closed Loop Control Ventilation | Manual Control Ventilation | Total
Number analyzed (Participants) | 104 | 102 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (13.07) | 39.6 (14.19) | 38.4 (13.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 82 | 79 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 27
  Not Hispanic or Latino | 88 | 86 | 174
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 22 | 48
  White | 65 | 67 | 132
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 10 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 104 | 102 | 206

OUTCOME MEASURES:

1. Primary Outcome: Relative Duration With Oxygen Saturation (SpO2) Within Target Range [Time Frame: 12 Hours]
Description: Relative duration is (time within SpO2 target of 92-96%)/12 hours where higher value demonstrates better ability of FiO2 control method to maintain appropriate oxygen saturation.
  Relative time the patient's SpO2 was maintained within target over the 12 hours on the study device, calculated as total time each patient had SpO2 within the 92 - 96% range divided by 12 hours with arcsin square root transformation
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Closed Loop Control Ventilation | Manual Control Ventilation
Number analyzed (Participants) | 104 | 102
arbitrary units | 0.53 (0.37) | 0.61 (0.36)

2. Primary Outcome: Number of Participants With SpO2 Less Than 88% at Anytime While on Study Device
Description: Number of participants with SpO2 less than 88% at anytime while on study device
Time Frame: 24 hours after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control Ventilation | Manual Control Ventilation
Number analyzed (Participants) | 104 | 102
Participants | 31 | 49

3. Secondary Outcome: Relative Duration of Time With SpO2 92 to 96% When FiO2 is Greater Than 21% and SpO2 is Greater Than or Equal to 92% When Fi02 "Relative Duration With Oxygen Saturation (SpO2) Within Target Range [Time Frame: 12 Hours]
Description: Relative duration is (time within SpO2 target of either a) 92-96% when FiO2 is greater than 21% or b) greater than or equal to 92% when FiO2 equals 21%)/12 hours where higher value demonstrates better ability of FiO2 control method to maintain appropriate oxygen saturation.
  Relative time the patient's SpO2 was maintained within target over the 12 hours on the study device, calculated as total time each patient had SpO2 within the range divided by 12 hours with arcsin square root transformation
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Closed Loop Control Ventilation | Manual Control Ventilation
Number analyzed (Participants) | 104 | 102
arbitrary units | 0.92 (0.34) | 0.83 (0.36)

ADVERSE EVENTS:
Time Frame: From enrollment until 24 hours after study device discontinuation, a period of 36 to 48 hours after study device placement.
Arm/Group | Closed Loop Control Ventilation | Manual Control Ventilation
All-Cause Mortality (participants affected / at risk) | 0/104 | 2/102
Serious Adverse Events (participants affected / at risk) | 0/104 | 9/102
Other Adverse Events (participants affected / at risk) | 24/104 | 17/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Closed Loop Control Ventilation (N=104) | Manual Control Ventilation (N=102)
Acute Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 0 | 1
Cerebral Edema (Nervous system disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Intracerbral hemorrhage (Nervous system disorders) | 0 | 1
Multi organ failure (General disorders) | 0 | 1
Pericardial Tamponade (Cardiac disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Subarachnoid hemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Closed Loop Control Ventilation (N=104) | Manual Control Ventilation (N=102)
Agitation (General disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bacteremia (Infections and infestations) | 0 | 1
Clostridium Difficle Infection (Infections and infestations) | 0 | 1
Coffee ground emesis (Gastrointestinal disorders) | 1 | 0
Device removal failed (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fever (Infections and infestations) | 3 | 4
gastric dilation (Gastrointestinal disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperoxemia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Hypovolemia (Vascular disorders) | 0 | 1
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Leukocytosis (Immune system disorders) | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mental status change (Nervous system disorders) | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 1
Neurological examination abnormal (Nervous system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Premature ventricular contractions (Cardiac disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Renal replacement therapy (Renal and urinary disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Swelling of eyelid (Eye disorders) | 1 | 0
Troponin increase (Cardiac disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT02810080/Prot_SAP_000.pdf